CLINICAL TRIAL: NCT01596335
Title: To Evaluate the Efficacy and Safety of TA-650 in Comparison With a Control Drug Polyethylene Glycol-treated Human Immunoglobulin (VGIH) in Patients With Kawasaki Disease Refractory to Initial Therapy With Intravenous Immunoglobulin (IVIG).
Brief Title: Clinical Study of TA-650 in Patients With Refractory Kawasaki Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-650-22
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Kawasaki Disease Refractory to Initial Therapy With Intravenous Immunoglobulin
Keywords: Infliximab; REMICADE; TA-650; intravenous immunoglobulin; Kawasaki disease; IVIG
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TA-650 (Experimental)
  Interventions: Drug: TA-650
- VGIH (Active Comparator)
  Interventions: Drug: Polyethylene Glycol-treated Human Immunoglobulin (VGIH)

INTERVENTIONS:
Drug: TA-650 — TA-650 at 5 mg per kg body weight on the day of TA-650 administration (day 0) is administered by intravenous infusion slowly over at least 2 hours.
  Arms: TA-650
Drug: Polyethylene Glycol-treated Human Immunoglobulin (VGIH) — VGIH at 2 g per kg body weight on the day of VGIH administration (day 0) is administered by intravenous infusion slowly over at least 20 hours.
  Arms: VGIH

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TA-650 in comparison with a control drug Polyethylene Glycol-treated Human Immunoglobulin (VGIH) in patients with Kawasaki disease refractory to initial therapy with Intravenous Immunoglobulin (IVIG). The pharmacokinetics of TA-650 is also examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Kawasaki disease (incipient cases only) with 5 or more of the 6 major symptoms of Kawasaki disease.
* Patients refractory to initial IVIG therapy (a single administration at 2 g per kg body weight).
* Patients with a fever of 37.5ºC or higher axillary temperature at the time of enrollment.
* Patients to whom the study drug can be administered by day 8 of disease.

Exclusion Criteria:

* Patients who have received vaccination with Bacille Calmette-Guérin (BCG) vaccine within 6 months before the enrollment.
* Patients with a complication, or a history within 6 months before the enrollment of, serious infections requiring hospitalization.
* Patients with a complication, or a history within 6 months before the enrollment of, opportunistic infections.
* Patients complicated with active tuberculosis, active hepatitis B or C, or patients confirmed to be hepatitis B virus carriers or a history of hepatitis B.
* Patients confirmed to have HIV infection, or patients with a family history of HIV infection.
* Patients who have a history of receiving treatment with infliximab or other biological products.
* Patients who had participated in another clinical study and had received a study drug within 12 weeks before giving consent.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Mori, MD, Study Director — Yokohama City University Medical Center
Locations (8):
- Japan (8):
  - Investigational site, Chugoku
  - Investigational site, Chūbu
  - Investigational site, Hokkaido
  - Investigational site, Kanto
  - Investigational site, Kyushu
  - Investigational site, Shinetu
  - Investigational site, Tōhoku
  - Investigational site, Tōkai

REFERENCES:
- [Result] Mori M, Hara T, Kikuchi M, Shimizu H, Miyamoto T, Iwashima S, Oonishi T, Hashimoto K, Kobayashi N, Waki K, Suzuki Y, Otsubo Y, Yamada H, Ishikawa C, Kato T, Fuse S. Infliximab versus intravenous immunoglobulin for refractory Kawasaki disease: a phase 3, randomized, open-label, active-controlled, parallel-group, multicenter trial. Sci Rep. 2018 Jan 31;8(1):1994. doi: 10.1038/s41598-017-18387-7. PMID 29386515

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyethylene Glycol-treated Human Immunoglobulin (VGIH): Polyethylene Glycol-treated Human Immunoglobulin (VGIH) at 2g per kg body weight on the day of VGIH administration (day 0) is administered by intravenous infusion slowly over at least 20 hours.
Period: Overall Study
Arm/Group | TA-650 | Polyethylene Glycol-treated Human Immunoglobulin (VGIH)
Started | 16 | 15
Completed | 11 | 6
Not Completed | 5 | 9
Not completed — exacerbation of primary disease | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TA-650 | Polyethylene Glycol-treated Human Immunoglobulin (VGIH) | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Customized [Number; unit: participants]
  >= 1 and < 2 | 2 | 2 | 4
  >= 2 and <= 10 | 14 | 13 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Defervescence Rate Within 48 Hours After the Start of the Study Drug Administration
Time Frame: Up to 48hours
Measure: Number; unit: percentage of patients
Arm/Group | TA-650 | Polyethylene Glycol-treated Human Immunoglobulin (VGIH)
Number analyzed (Participants) | 16 | 15
percentage of patients | 75.0 | 33.3

2. Secondary Outcome: Duration of Fever
Time Frame: Up to Day56
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | TA-650 | Polyethylene Glycol-treated Human Immunoglobulin (VGIH)
Number analyzed (Participants) | 16 | 15
hour
  Duration since starting of drug administration | 16.00 [7.70 to 38.75] | 42.20 [20.00 to 60.70]
  Duration since completing of drug administration | 13.90 [5.90 to 36.50] | 25.90 [17.30 to 39.80]

3. Secondary Outcome: Incidence of Coronary Artery Lesions
Time Frame: Day 3, Day 7, Day14, Day 21, Day56
Population: The analysis population is evaluation patients.
Measure: Number; unit: percentage of patients
Arm/Group | TA-650 | Polyethylene Glycol-treated Human Immunoglobulin (VGIH)
Number analyzed (Participants) | 16 | 15
percentage of patients
  Day 3: number analyzed (Participants) | 13 | 8
  Day 3 | 0 | 12.5
  Day 7: number analyzed (Participants) | 13 | 7
  Day 7 | 0 | 14.3
  Day14: number analyzed (Participants) | 12 | 6
  Day14 | 0 | 16.7
  Day 21: number analyzed (Participants) | 11 | 5
  Day 21 | 0 | 20.0
  Day56: number analyzed (Participants) | 11 | 6
  Day56 | 0 | 0.0

ADVERSE EVENTS:
Arm/Group | TA-650 | Polyethylene Glycol-treated Human Immunoglobulin (VGIH)
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/15
Other Adverse Events (participants affected / at risk) | 15/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=16) | Polyethylene Glycol-treated Human Immunoglobulin (VGIH) (N=15)
Kawasaki disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=16) | Polyethylene Glycol-treated Human Immunoglobulin (VGIH) (N=15)
Bronchitis (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Neuralgia (Nervous system disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Disuse syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Double stranded DNA antibody positive (Investigations) | 11 | 10
Eosinophil count increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other